CLINICAL TRIAL: NCT01772615
Title: Active Ulcerative Colitis; Placebo Controlled Treatment Trial With Ciprofloxacin and E. Coli Nissle
Brief Title: Treatment of Ulcerative Colitis With Ciprofloxacin and E. Coli Nissle
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Andreas Munk Petersen, MD, ph.d., Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-1-2009-10
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Ulcerative Colitis
Keywords: EcN, Nissle, Mutaflor, Ulcerative Colitis, antibiotics, Inflammatory Bowel Diseases
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ciprofloxacin-EcN (Experimental)
  Interventions: Drug: Ciprofloxacin; Dietary Supplement: E. coli Nissle
- ciprofloxacin-placebo (Experimental)
  Interventions: Drug: Ciprofloxacin
- placebo-EcN (Experimental)
  Interventions: Dietary Supplement: E. coli Nissle
- placebo-placebo (Placebo Comparator)

INTERVENTIONS:
Drug: Ciprofloxacin — Antibiotic
  Arms: ciprofloxacin-EcN; ciprofloxacin-placebo
Dietary Supplement: E. coli Nissle — Probiotic
  Arms: ciprofloxacin-EcN; placebo-EcN

SUMMARY:
Purpose: The purpose of the study is to investigate if treatment with ciprofloxacin for one week followed by therapy with E. Coli Nissle (EcN) for seven weeks can influence disease activity among ulcerative colitis patients with disease flare-ups compared to placebo controls.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic inflammatory bowel disease where existing treatments have proven to result in numerous side effects. An important causal factor for the development of the disease is an autoimmune cellular response against bacteria in the colon.

As a possible treatment, manipulation of the bacterial flora has been studied using the probiotic bacterium Escherichia coli Nissle 1917 (EcN). Studies on UC patients have shown that treatment with EcN is equally good at maintaining remission as the standard treatment with mesalazine. Furthermore, treatment with antibiotics such as ciprofloxacin have been studied for treatment of UC and some, but shortlived, effect has been described.

Patients are randomized to one of four treatment-arms: ciprofloxacin-EcN, ciprofloxacin-placebo, placebo-EcN or placebo-placebo.

Disease activity are quantitated with Colitis Activity Index (CAI) and quality of life by the Inflammatory Bowel Disease Questionnaire (IBDQ). Also, dietary interviews to examine the patients' dietary intake are completed and the patients' fecal-calprotectin-concentrations will be measured.

Hundred subjects with ulcerative colitis will be recruited for the study. Standard medical care and therapies will be continued throughout the study

ELIGIBILITY:
Inclusion Criteria:

* Age, >/=18 years and diagnosed with ulcerative colitis
* CAI score of >/=6 (active UC)

Exclusion Criteria:

* Pregnant or breastfeeding females
* Known sensitivity to ciprofloxacin
* Subjects who participate in another clinical trial
* Positive stool sample with any enteric pathogens, parasites or Clostridium difficile
* Treatment with systemic corticosteroids or biologic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Compare number of participants in remission | 12 weeks
  Compare number of participants in remission (CAI </=4) in the four groups. Compare time to the patients achieve remission (CAI </=4) in the four groups

SECONDARY OUTCOMES:
Compare numbers of patients who completed the study in the 4 groups | 12 weeks
  Compare numbers of patients who completed the study in the 4 groups Compare IBDQ-score in the 4 groups Compare dietary intake in the 4 groups Compare the possible side effects of treatment in the different groups

OTHER OUTCOMES:
E. coli strains | 12 weeks
  Compare changes in E. coli strains in the 4 groups

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Petersen, MD, ph.d., Principal Investigator — Hvidovre University Hospital; Andreas M Petersen, MD, ph.d., Study Chair — Hvidovre University Hospital
Locations (1):
- Hvidovre Hospital, Copenhagen University, Hvidovre, Copenhagen, Denmark

REFERENCES:
- [Background] Vejborg RM, Hancock V, Petersen AM, Krogfelt KA, Klemm P. Comparative genomics of Escherichia coli isolated from patients with inflammatory bowel disease. BMC Genomics. 2011 Jun 15;12:316. doi: 10.1186/1471-2164-12-316. PMID 21676223
- [Background] Petersen AM, Nielsen EM, Litrup E, Brynskov J, Mirsepasi H, Krogfelt KA. A phylogenetic group of Escherichia coli associated with active left-sided inflammatory bowel disease. BMC Microbiol. 2009 Aug 20;9:171. doi: 10.1186/1471-2180-9-171. PMID 19695087
- See also: Related Info — http://www.ssi.dk/Service/Sygdomsleksikon/C/~/media/Indhold/DK%20-%20dansk/Sygdomsleksikon/colitis%20ulcerosaE%20coli%20Nissle%20projekt.ashx